CLINICAL TRIAL: NCT06828146
Title: A Quasi-Experimental Study on Developing Social Justice Advocacy in Nursing Education Through Critical Pedagogy and Freirean Dialogues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, FUNDA ASLAN, Assist.Prof., Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAKU-01-10-2024
Record Dates: First submitted 2025-02-09; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Social Justice Advocacy; Nursing Education

STUDY DESIGN:
Intervention Model Description: This study employs a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dia (Experimental): a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.
  Interventions: Other: a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.

INTERVENTIONS:
Other: a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students. — a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.

SUMMARY:
Recognizing the critical significance of social and health inequalities as one of the foremost global challenges, the United Nations (UN) acknowledged the growing disparity as a key issue in the Millennium Development Goals (MDG). Reducing global inequalities was established as one of the 17 MDG targets for the period 2015-2030. While certain health indicators have seen improvement in Turkey's healthcare system, notable factors continue to threaten the equitable provision of healthcare. In light of the profound societal transformations in Turkey, including a substantial influx of refugees and ongoing economic challenges, the pursuit of social justice has become essential (Makovsky, 2019). Therefore, it is crucial to position social justice as a central theme in nursing education (Einhellig et al., 2016; Hellman et al., 2018). Nevertheless, scholarly literature highlights the importance of exploring how nurse educators can foster this comprehension and motivate students towards the aim of advocacy. The literature underscores the dual significance of addressing this topic in nursing education (Hellman et al., 2018), while also emphasizing the need to broaden understanding of effective teaching and learning strategies. These methods are essential for equipping students with the knowledge and skills necessary to advocate for social justice, empowering them to critically examine existing systems, develop a sense of agency, and take responsibility for driving societal change in nursing practice (Elliott & Sandberg, 2021).

Historically, nursing education has operated within a culture of silence, often neglecting issues of oppression, racism, and marginalization. This stands in contrast to Freire's Pedagogy of the Oppressed, which emphasizes dialogue as a fundamental element of teaching and learning (Iheduru-Anderson et al., 2021, 2022). By incorporating dialogical methods in nursing classrooms, educators can create inclusive spaces where students openly share their experiences, engage in meaningful discussions on social justice, and collaborate in knowledge creation. Such reciprocal dialogue is only possible in environments that value diverse perspectives and foster a sense of belonging (Kechi et al., 2024) Through dialogical education, students gain confidence, actively participate in their learning, and develop the critical thinking skills necessary to challenge inequities (Giroux, 2010; Paulo Freire et al., 2014). Integrating Freire's critical pedagogy into nursing education not only strengthens these skills but also prepares nurses to advocate for social change, ultimately contributing to a more just and equitable healthcare system (Kechi et al., 2024). The current study applies Paulo Freire's critical pedagogy, highlighting education as a means of empowerment and encouraging learners to critically analyze societal structures while engaging in transformative action. Integrating Freirean principles can cultivate critical consciousness among students, equipping them to identify and address systemic inequalities in healthcare.

This study employs a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.

DETAILED DESCRIPTION:
Social justice, deeply rooted in nursing history, is best understood as both a process and an outcome, encompassing attributes such as fairness, justness, equity, and well-being (Thurman & Pfitzinger-Lippe, 2017). There is a global consensus that social justice is intrinsically linked to health and health equity, making it highly pertinent for nursing education.

From the perspective of nursing care, There is pre-pandemic evidence on the barriers to this important contribution to global health, including being a female predominant workforce and has long faced barriers to effective advocacy, based on the gendered identity (Madigan et al., 2023) The COVID-19 pandemic underscored nurses are important advocates for the world's population. Numerous studies have highlighted that the pandemic has worsened health disparities, emphasizing the crucial role of nurses in conducting health promotion and disease prevention efforts for the global population After the pandemic, The World Health Organization (WHO) reports that the detrimental impacts of socioeconomic inequalities are increasingly evident in today's societies. In response to these findings, the International Council of Nurses (ICN) emphasizes strongly that nurses are professionally obligated to champion equity and social justice (ICN, 2023) They have a responsibility for initiating and backing actions aimed at addressing the health and social needs of the public, especially those belonging to vulnerable populations. The urgency for nurses to advocate for equity and social justice is intensifying with each day, as societal and healthcare disparities continue to evolve and become more apparent.

Despite the growing need to cultivate a healthcare workforce equipped to address social injustice in practical settings. There's a scarcity of research exploring the integration of social justice into undergraduate nursing education (Einhellig et al., 2016; Habibzadeh et al., 2021; Houston et al., 2023; Roy et al., 2022; Shahzad et al., 2022) A study conducted in Iran revealed that inadequate focus on social justice within educational settings hampers nurses' ability to contribute to the establishment of social justice within the healthcare system (Hosseinzadegan et al., 2021). Habibzadeh et al. (2021) demonstrated significant shortcomings in teaching the concept of social justice within nursing education and They underscored the imperative need to revise the content of nursing curricula and educational methodologies to effectively instill this fundamental value. Valderama-Wallace and Apesoa-Varano (2019) noted that nurse educators express concerns regarding their limited endeavors to enhance this foundational value. Additionally, they highlighted a lack of structural and institutional support for such efforts. Two reviews conducted in 2022 and 2023 uncovered a deficiency in research dedicated to improving social justice within nursing education, with a significant portion of the studies originating from the USA (Abu & Moorley, 2023; Shahzad et al., 2022). This underscores the importance of nursing schools in the European region and other countries facing challenges such as hosting refugees and grappling with social and economic issues, need to prioritize the integration of social justice into undergraduate nursing education (Abu & Moorley, 2023; Valderama-Wallace & Apesoa-Varano, 2019)

Turkey is among the notable countries experiencing recent societal changes. As is widely recognized, the root of health disparities often lies in challenging socioeconomic circumstances, causing the most marginalized communities to consistently experience inferior health outcomes. In Turkey, societal shifts such as significant migration influxes and deteriorating socioeconomic conditions can serve as significant contributors to social injustice. Despite these concerns, regrettably, there remains a substantial gap concerning social justice issues within the Turkish nursing education system. Only one study has utilized the nursing education curriculum to enhance social justice advocacy among nursing students. Nonetheless, Turkish educators must enhance social justice in nursing education by employing various methods.

Traditional lecture formats offer limited advantages in conveying abstract concepts like social justice. Given the demands of nursing professional roles, students must start evaluating their moral framework, equipping them to effectively care for and advocate for diverse patient populations. To effectively convey this crucial concept to nursing students, nursing faculty must employ diverse pedagogical strategies (Einhellig et al., 2016). These strategies may deepen their awareness of social inequality from alternative perspectives, thereby framing the significance of taking action in the face of social injustice within healthcare settings.

Paulo Freire's critical pedagogy is an educational approach that emphasizes the transformative power of education in challenging and dismantling oppressive societal structures (Paulo Freire et al., 2014) At its core, this pedagogy prioritizes dialogue, framing education as a means of liberation by encouraging learners to critically examine their realities and take action for change (Giroux, 2010; Paulo Freire et al., 2014).

Applying Freire's principles in education involves fostering a learning environment that promotes critical reflection, open dialogue, and active engagement. This approach empowers students to question existing systems, cultivate a sense of agency, and take responsibility for societal transformation (Rozendo et al., 2017).

Historically, nursing education has operated within a culture of silence, often neglecting issues of oppression, racism, and marginalization. This stands in contrast to Freire's Pedagogy of the Oppressed, which emphasizes dialogue as a fundamental element of teaching and learning (Iheduru-Anderson et al., 2021, 2022). By incorporating dialogical methods in nursing classrooms, educators can create inclusive spaces where students openly share their experiences, engage in meaningful discussions on social justice, and collaborate in knowledge creation. Such reciprocal dialogue is only possible in environments that value diverse perspectives and foster a sense of belonging (Kechi et al., 2024) Through dialogical education, students gain confidence, actively participate in their learning, and develop the critical thinking skills necessary to challenge inequities (Giroux, 2010; Paulo Freire et al., 2014). Integrating Freire's critical pedagogy into nursing education not only strengthens these skills but also prepares nurses to advocate for social change, ultimately contributing to a more just and equitable healthcare system (Kechi et al., 2024). The current study applies Paulo Freire's critical pedagogy, highlighting education as a means of empowerment and encouraging learners to critically analyze societal structures while engaging in transformative action. Integrating Freirean principles can cultivate critical consciousness among students, equipping them to identify and address systemic inequalities in healthcare.

Method This study employs a quasi-experimental one-group pretest-posttest design to evaluate the effectiveness of Freirean dialogue-based critical pedagogy in fostering social justice advocacy among nursing students.

Participants Population: Undergraduate nursing students from a Turkish nursing school. Sample Size: 85 students were recruited through purposive sampling.

Procedure

The six-week intervention consisted of:

Critical Reflection Sessions: Students engaged in structured discussions on healthcare inequities.

Problem-Posing Learning: case studies on marginalized populations and healthcare discrimination.

Freirean Dialogues: Student-led discussions focusing on social determinants of health

ELIGIBILITY:
Inclusion Criteria:

Nursing students enrolled in nursing ethics courses. No prior formal training in social justice advocacy

Exclusion Criteria:

Students with previous participation in social justice-related workshops or courses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
pirmary outcome | 6 weeks
  • Higher posttest scores compared to pretest, indicating improved advocacy knowledge, confidence, and engagement

CONTACTS AND LOCATIONS:
Locations (1):
- Cankırı Karatekin University, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paulo Freire, Myra Bergman Ramos, & Myra Bergman Ramos. (2014). Pedagogy_of_the_Oppressed_30th_Anniversary_Edition_----_(Chapter_4). In Pedagogy of the Oppressed: 30th Anniversary Edition (pp. 125-185).
- [Background] Kechi IA, Waite R, Murray TA. Examining and mitigating racism in nursing using the socio-ecological model. Nurs Inq. 2024 Jul;31(3):e12639. doi: 10.1111/nin.12639. Epub 2024 Apr 3. PMID 38567694
- [Background] Iheduru-Anderson K, Okoro FO, Moore SS. Diversity and Inclusion or Tokens? A Qualitative Study of Black Women Academic Nurse Leaders in the United States. Glob Qual Nurs Res. 2022 Jan 18;9:23333936211073116. doi: 10.1177/23333936211073116. eCollection 2022 Jan-Dec. PMID 35097160
- [Background] Giroux, H. A. (2010). Rethinking education as the practice of freedom: Paulo Freire and the promise of critical pedagogy. Policy Futures in Education, 8(6), 715-721. https://doi.org/10.2304/pfie.2010.8.6.715